CLINICAL TRIAL: NCT07138872
Title: The Effect of Surgical Position on Hemodynamics in Percutaneous Nephrolithotomy Performed in Prone and Supine Positions
Brief Title: Hemodynamic Effects of Surgical Position in Prone vs. Supine Percutaneous Nephrolithotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Arif Burak Keçebaş, UROLOGY DOCTOR, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-SBF-ABK-01
Record Dates: First submitted 2025-08-09; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Percutaneous Nephrolithotomy (PCNL); Surgical Positioning; Prone Position; Supine Position; Hemodynamic Stability; Nephrolithiasis
Keywords: PCNL; Prone Position; Percutaneous Nephrolithotomy; Supine Position; Hemodynamic stability; Nephrolithiasis
MeSH Terms: conditions — Deception; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Position (Experimental): Patients in this group will undergo percutaneous nephrolithotomy (PNL) in the prone position. The procedure begins with ureteral catheter placement in lithotomy position, followed by prone positioning for renal access under C-arm fluoroscopic guidance. Stone fragmentation will be performed using pneumatic or ultrasonic lithotripters, and nephrostomy placement will be completed according to standard protocol.
  Interventions: Procedure: Prone Position Percutaneous Nephrolithotomy
- Supine Position (Experimental): Patients in this group will undergo percutaneous nephrolithotomy (PNL) in the Galdakao-modified Valdivia supine position. Following general anesthesia, the ipsilateral side will be elevated 20-30°, with the ipsilateral leg extended and the contralateral leg abducted. Ureteral catheter placement will be followed by renal access under C-arm fluoroscopy. Stone fragmentation and removal will be performed using the same standardized lithotripsy and irrigation protocols as in the prone group.
  Interventions: Procedure: Supine Position Percutaneous Nephrolithotomy (Galdakao-modified Valdivia)

INTERVENTIONS:
Procedure: Prone Position Percutaneous Nephrolithotomy — Patients in this arm will undergo percutaneous nephrolithotomy (PNL) in the prone position. The procedure begins with ureteral catheter placement in lithotomy position, followed by prone positioning for renal access under C-arm fluoroscopic guidance. Stone fragmentation will be performed using pneumatic or ultrasonic lithotripters, and nephrostomy placement will be completed according to standard protocol.
  Arms: Prone Position
Procedure: Supine Position Percutaneous Nephrolithotomy (Galdakao-modified Valdivia) — Patients in this arm will undergo percutaneous nephrolithotomy (PNL) in the Galdakao-modified Valdivia supine position. Following general anesthesia, the ipsilateral side will be elevated 20-30°, with the ipsilateral leg extended and the contralateral leg abducted. Ureteral catheter placement will be followed by renal access under C-arm fluoroscopy. Stone fragmentation and removal will be performed using the same standardized lithotripsy and irrigation protocols as in the prone group.
  Arms: Supine Position

SUMMARY:
This prospective, randomized controlled study evaluates the hemodynamic effects of prone and supine positions during percutaneous nephrolithotomy (PNL) for large kidney stones. Surgical position may influence intraoperative and postoperative hemodynamic stability. Prone positioning can increase intrathoracic pressure and reduce venous return, whereas supine positioning may provide greater hemodynamic stability. A total of 84 patients will be randomized to undergo PNL in prone or supine positions. Primary outcomes include changes in hemodynamic parameters during surgery. Results may guide surgical position selection, especially in patients with potential hemodynamic risk.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PNL) is a widely used minimally invasive surgical technique for the treatment of large and complex renal calculi. Traditionally, PNL has been performed in the prone position; however, the supine position has gained popularity in recent years due to potential anesthetic and surgical advantages. Surgical positioning can significantly influence cardiovascular and respiratory function, potentially leading to intraoperative and postoperative hemodynamic fluctuations.

Previous literature suggests that the prone position may increase intrathoracic pressure and impair venous return, potentially compromising hemodynamic stability, while the supine position may provide a more stable cardiovascular profile. However, existing data are limited, and results remain inconclusive, particularly in direct comparative studies.

This prospective, randomized controlled clinical trial aims to compare the effects of prone and supine positions during PNL on patients' intraoperative and postoperative hemodynamic parameters. The study will enroll 84 patients aged 18-80 years with American Society of Anesthesiologists (ASA) physical status I-III undergoing elective PNL. Patients will be randomly assigned to either the prone (n=42) or supine (n=42) position.

Inclusion criteria include patients with renal calculi suitable for PNL and meeting the study's eligibility requirements. Exclusion criteria include pregnancy, uncontrolled coagulopathy, previous renal surgery, severe cardiac, pulmonary, or neurological disease, preoperative urinary tract infection, surgery duration outside 60-120 minutes, and multiple access tracts.

Preoperative evaluation will include demographic data, stone characteristics, and relevant laboratory and imaging findings. Intraoperative data will include systolic and diastolic blood pressure, heart rate, arterial blood gas analysis, operative time, anesthesia duration, access details, irrigation volume, and any transfusion or complications. Postoperative parameters will include nephrostomy duration, length of hospital stay, and presence of residual stones as assessed by postoperative CT scan.

Surgical techniques will be standardized for both positions. Prone PNL will involve initial lithotomy positioning for ureteral catheter placement followed by prone positioning for renal access under fluoroscopic guidance. Supine PNL will be performed in the Galdakao-modified Valdivia position with similar access and fragmentation protocols.

The primary outcome is the difference in intraoperative and postoperative hemodynamic stability between positions. Secondary outcomes include complication rates, residual stone rates, and hospital stay duration.

This study aims to provide high-quality evidence to guide surgeons and anesthesiologists in selecting the optimal patient position for PNL, particularly in individuals with higher hemodynamic risk.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* Presence of renal calculi indicated for PNL

Exclusion Criteria:

* Pregnancy
* Uncontrolled coagulopathy
* Previous renal surgery
* Severe cardiac, pulmonary, or neurological disease
* Preoperative urinary tract infection (non-sterile urine culture)
* Surgery duration <60 minutes or >120 minutes
* Preoperative blood transfusion
* Multiple access tracts

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hemodynamic Parameters (Intraoperative) | From induction of anesthesia to the end of surgery (approximately 60-120 minutes)
  Systolic blood pressure (mmHg) will be recorded at predefined time points (preoperative baseline, intraoperative intervals, and immediate postoperative period) to assess intraoperative hemodynamic stability.
Change in Arterial Blood pH | Preoperative, intraoperative, postoperative day 1
  Arterial pH will be measured at predefined time points (preoperative, intraoperative, postoperative day 1) to evaluate metabolic changes between prone and supine groups.
Change in Diastolic Blood Pressure (Intraoperative) | From induction of anesthesia to the end of surgery (approximately 60-120 minutes
  Diastolic blood pressure (mmHg) will be recorded at predefined time points (preoperative baseline, intraoperative intervals, and immediate postoperative period) to assess intraoperative hemodynamic stability.
Change in Mean Arterial Pressure (Intraoperative) | From induction of anesthesia to the end of surgery (approximately 60-120 minutes)
  Mean arterial pressure (mmHg) will be recorded at predefined time points (preoperative baseline, intraoperative intervals, and immediate postoperative period) to assess intraoperative hemodynamic stability.
Change in Heart Rate (Intraoperative) | From induction of anesthesia to the end of surgery (approximately 60-120 minutes)
  Heart rate (beats per minute) will be recorded at predefined time points (preoperative baseline, intraoperative intervals, and immediate postoperative period) to assess intraoperative hemodynamic stability.
Change in Arterial pO₂ | Preoperative, intraoperative, postoperative day 1
  Arterial oxygen partial pressure (mmHg) will be measured at predefined time points (preoperative, intraoperative, postoperative day 1) to evaluate respiratory function.
Change in Arterial HCO₃- | Preoperative, intraoperative, postoperative day 1
  Arterial bicarbonate (mmol/L) will be measured at predefined time points (preoperative, intraoperative, postoperative day 1) to evaluate metabolic changes.
Change in Oxygen Saturation | Preoperative, intraoperative, postoperative day 1
  Arterial oxygen saturation (%) will be measured at predefined time points (preoperative, intraoperative, postoperative day 1) to evaluate respiratory status.
Change in Arterial pCO₂ | Preoperative, intraoperative, postoperative day 1
  Arterial carbon dioxide partial pressure (mmHg) will be measured at predefined time points (preoperative, intraoperative, postoperative day 1) to evaluate respiratory changes.

SECONDARY OUTCOMES:
Operative Time | From initial skin incision until completion of stone removal (approximately 30-180 minutes).
  Total time from initial skin incision to completion of stone removal will be recorded for each group.
Anesthesia Duration | From induction of anesthesia until termination of anesthesia and awakening of the patient (approximately 60-240 minutes).
  Total anesthesia time will be measured to assess any differences related to patient positioning.
Intraoperative Blood Loss | Intraoperative period (from skin incision to completion of surgery, approximately 30-180 minutes).
  Estimated blood loss will be calculated and recorded; intraoperative transfusion requirements will also be noted.
Complication Rate | From intraoperative period through hospital stay and up to 30 days postoperatively.
  Complications will be identified and classified according to the Clavien-Dindo classification system.
Residual Stone Rate | At postoperative 1 month, assessed by CT scan.
  Presence of residual stones larger than 4 mm will be recorded; stones ≤4 mm will be considered clinically insignificant.
Length of Hospital Stay | From hospital admission until discharge (typically 2-10 days).
  The total number of days of hospitalization will be compared between groups.
Nephrostomy Tube Duration | From postoperative day 0 (day of surgery) until nephrostomy tube removal, typically within 7-14 days.
  The duration (in days) that the nephrostomy tube remains in place will be recorded for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Arslan, CLINICAL PROFESSOR OF UROLOGY, Study Director — Gaziosmanpaşa Training and Research Hospital, Urology Department, Istanbul, Türkiye
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No